CLINICAL TRIAL: NCT04552405
Title: Preventive Anti-inflammatory Diet to Reduce Gastro-intestinal Inflammation in FAP Patients: a Prospective Pilot Study
Acronym: FAPPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: INT 78/17
Record Dates: First submitted 2020-05-04; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-05

CONDITIONS: Familial Adenomatous Polyposis (FAP)
Keywords: FAP; Familial Adenomatous Polyposis
MeSH Terms: conditions — Adenomatous Polyposis Coli

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAP patients (Other): FAP patients who underwent prophylactic total colectomy
  Interventions: Dietary Supplement: Anti-inflammatory Diet

INTERVENTIONS:
Dietary Supplement: Anti-inflammatory Diet — FAP individuals followed for 3 months a low-inflammatory diet

SUMMARY:
Preventive anti-inflammatory diet to reduce gastro-intestinal inflammation in FAP patients: a prospective pilot study

DETAILED DESCRIPTION:
a prospective pilot study

ELIGIBILITY:
Inclusion Criteria:

- FAP patients carrying mutations in APC gene, submitted to prophylactic total colectomy/IRA (with rectum preservation) and that participate to the regular endoscopic surveillance program at IRCCS-INT.

Exclusion Criteria:

* FAP patients taking NSAIDs and/or Omega 3
* Patients who carried MUTYH germline mutations or had no APC mutation found.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
Evaluate changes in calprotectin levels | baseline, at 3 months and 6 months post anti-inflammatory diet consumption.
  Change from baseline in calprotectin levels at 3 months and 6 months post anti-inflammatory diet consumption.

SECONDARY OUTCOMES:
Evaluate changes in circulatory inflammatory markers | baseline, at 3 months and 6 months post anti-inflammatory diet consumption.
  Change from baseline in circulatory inflammatory markers at 3 months and 6 months post anti-inflammatory diet consumption.
Evaluate the effect on polyps growth | baseline and 6 months post anti-inflammatory diet consumption
  Evaluate the effect of the anti-inflammatory diet on polyps growth in the rectal stump (in terms of number of polyps)
Evaluate changes in the number of diarrheal discharges | baseline, at 3 months and 6 months post anti-inflammatory diet consumption
  Change from baseline in the number of diarrheal discharges at 3 months and 6 months post anti-inflammatory diet consumption
Evaluate changes in the immune cell profile | baseline, at 3 months and 6 months post anti-inflammatory diet consumption
  Change from baseline in the immune cell profile at 3 months and 6 months post anti-inflammatory diet consumption
Evaluate changes in stool inflammatory markers | baseline, at 3 months and 6 months post anti-inflammatory diet consumption
  Change from baseline in stool inflammatory markers at 3 months and 6 months post anti-inflammatory diet consumption

CONTACTS AND LOCATIONS:
Overall Officials: Marco Vitellaro, MD, Principal Investigator — Fondazione IRCCS ISTITUTO NAZIONALE TUMORI
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
It will be discussed later by the staff

REFERENCES:
- [Background] Vasen HF, Moslein G, Alonso A, Aretz S, Bernstein I, Bertario L, Blanco I, Bulow S, Burn J, Capella G, Colas C, Engel C, Frayling I, Friedl W, Hes FJ, Hodgson S, Jarvinen H, Mecklin JP, Moller P, Myrhoi T, Nagengast FM, Parc Y, Phillips R, Clark SK, de Leon MP, Renkonen-Sinisalo L, Sampson JR, Stormorken A, Tejpar S, Thomas HJ, Wijnen J. Guidelines for the clinical management of familial adenomatous polyposis (FAP). Gut. 2008 May;57(5):704-13. doi: 10.1136/gut.2007.136127. Epub 2008 Jan 14. PMID 18194984
- [Background] Ullman TA, Itzkowitz SH. Intestinal inflammation and cancer. Gastroenterology. 2011 May;140(6):1807-16. doi: 10.1053/j.gastro.2011.01.057. PMID 21530747
- [Background] Giardiello FM, Hamilton SR, Krush AJ, Piantadosi S, Hylind LM, Celano P, Booker SV, Robinson CR, Offerhaus GJ. Treatment of colonic and rectal adenomas with sulindac in familial adenomatous polyposis. N Engl J Med. 1993 May 6;328(18):1313-6. doi: 10.1056/NEJM199305063281805. PMID 8385741
- [Background] Dolan KT, Chang EB. Diet, gut microbes, and the pathogenesis of inflammatory bowel diseases. Mol Nutr Food Res. 2017 Jan;61(1):10.1002/mnfr.201600129. doi: 10.1002/mnfr.201600129. Epub 2016 Aug 15. PMID 27346644
- [Background] Neuhouser ML, Schwarz Y, Wang C, Breymeyer K, Coronado G, Wang CY, Noar K, Song X, Lampe JW. A low-glycemic load diet reduces serum C-reactive protein and modestly increases adiponectin in overweight and obese adults. J Nutr. 2012 Feb;142(2):369-74. doi: 10.3945/jn.111.149807. Epub 2011 Dec 21. PMID 22190020
- [Background] Esmaillzadeh A, Kimiagar M, Mehrabi Y, Azadbakht L, Hu FB, Willett WC. Fruit and vegetable intakes, C-reactive protein, and the metabolic syndrome. Am J Clin Nutr. 2006 Dec;84(6):1489-97. doi: 10.1093/ajcn/84.6.1489. PMID 17158434
- [Background] Azadbakht L, Esmaillzadeh A. Red meat intake is associated with metabolic syndrome and the plasma C-reactive protein concentration in women. J Nutr. 2009 Feb;139(2):335-9. doi: 10.3945/jn.108.096297. Epub 2008 Dec 11. PMID 19074209
- [Background] Esmaillzadeh A, Azadbakht L. Home use of vegetable oils, markers of systemic inflammation, and endothelial dysfunction among women. Am J Clin Nutr. 2008 Oct;88(4):913-21. doi: 10.1093/ajcn/88.4.913. PMID 18842776
- [Background] Azadbakht L, Kimiagar M, Mehrabi Y, Esmaillzadeh A, Hu FB, Willett WC. Soy consumption, markers of inflammation, and endothelial function: a cross-over study in postmenopausal women with the metabolic syndrome. Diabetes Care. 2007 Apr;30(4):967-73. doi: 10.2337/dc06-2126. PMID 17392557
- [Background] de Oliveira Otto MC, Alonso A, Lee DH, Delclos GL, Jenny NS, Jiang R, Lima JA, Symanski E, Jacobs DR Jr, Nettleton JA. Dietary micronutrient intakes are associated with markers of inflammation but not with markers of subclinical atherosclerosis. J Nutr. 2011 Aug;141(8):1508-15. doi: 10.3945/jn.111.138115. Epub 2011 Jun 8. PMID 21653577
- [Background] Flock MR, Rogers CJ, Prabhu KS, Kris-Etherton PM. Immunometabolic role of long-chain omega-3 fatty acids in obesity-induced inflammation. Diabetes Metab Res Rev. 2013 Sep;29(6):431-45. doi: 10.1002/dmrr.2414. PMID 23592441
- [Background] Rankin JW, Turpyn AD. Low carbohydrate, high fat diet increases C-reactive protein during weight loss. J Am Coll Nutr. 2007 Apr;26(2):163-9. doi: 10.1080/07315724.2007.10719598. PMID 17536128
- [Background] Fu Z, Shrubsole MJ, Smalley WE, Wu H, Chen Z, Shyr Y, Ness RM, Zheng W. Lifestyle factors and their combined impact on the risk of colorectal polyps. Am J Epidemiol. 2012 Nov 1;176(9):766-76. doi: 10.1093/aje/kws157. Epub 2012 Oct 18. PMID 23079606
- [Background] Olendzki BC, Silverstein TD, Persuitte GM, Ma Y, Baldwin KR, Cave D. An anti-inflammatory diet as treatment for inflammatory bowel disease: a case series report. Nutr J. 2014 Jan 16;13:5. doi: 10.1186/1475-2891-13-5. PMID 24428901
- [Background] Samadder NJ, Gornick M, Everett J, Greenson JK, Gruber SB. Inflammatory bowel disease and familial adenomatous polyposis. J Crohns Colitis. 2013 Apr;7(3):e103-7. doi: 10.1016/j.crohns.2012.06.021. Epub 2012 Jul 17. PMID 22809634
- [Background] Henson CC, Burden S, Davidson SE, Lal S. Nutritional interventions for reducing gastrointestinal toxicity in adults undergoing radical pelvic radiotherapy. Cochrane Database Syst Rev. 2013 Nov 26;2013(11):CD009896. doi: 10.1002/14651858.CD009896.pub2. PMID 24282062
- [Background] Chun E, Lavoie S, Michaud M, Gallini CA, Kim J, Soucy G, Odze R, Glickman JN, Garrett WS. CCL2 Promotes Colorectal Carcinogenesis by Enhancing Polymorphonuclear Myeloid-Derived Suppressor Cell Population and Function. Cell Rep. 2015 Jul 14;12(2):244-57. doi: 10.1016/j.celrep.2015.06.024. Epub 2015 Jul 2. PMID 26146082
- [Background] Dennis KL, Wang Y, Blatner NR, Wang S, Saadalla A, Trudeau E, Roers A, Weaver CT, Lee JJ, Gilbert JA, Chang EB, Khazaie K. Adenomatous polyps are driven by microbe-instigated focal inflammation and are controlled by IL-10-producing T cells. Cancer Res. 2013 Oct 1;73(19):5905-13. doi: 10.1158/0008-5472.CAN-13-1511. Epub 2013 Aug 16. PMID 23955389
- [Background] Mlecnik B, Bindea G, Angell HK, Maby P, Angelova M, Tougeron D, Church SE, Lafontaine L, Fischer M, Fredriksen T, Sasso M, Bilocq AM, Kirilovsky A, Obenauf AC, Hamieh M, Berger A, Bruneval P, Tuech JJ, Sabourin JC, Le Pessot F, Mauillon J, Rafii A, Laurent-Puig P, Speicher MR, Trajanoski Z, Michel P, Sesboue R, Frebourg T, Pages F, Valge-Archer V, Latouche JB, Galon J. Integrative Analyses of Colorectal Cancer Show Immunoscore Is a Stronger Predictor of Patient Survival Than Microsatellite Instability. Immunity. 2016 Mar 15;44(3):698-711. doi: 10.1016/j.immuni.2016.02.025. PMID 26982367
- [Background] Biswas SK. Metabolic Reprogramming of Immune Cells in Cancer Progression. Immunity. 2015 Sep 15;43(3):435-49. doi: 10.1016/j.immuni.2015.09.001. PMID 26377897
- [Background] Honda K, Littman DR. The microbiota in adaptive immune homeostasis and disease. Nature. 2016 Jul 7;535(7610):75-84. doi: 10.1038/nature18848. PMID 27383982
- [Background] Louis P, Hold GL, Flint HJ. The gut microbiota, bacterial metabolites and colorectal cancer. Nat Rev Microbiol. 2014 Oct;12(10):661-72. doi: 10.1038/nrmicro3344. Epub 2014 Sep 8. PMID 25198138
- [Background] Laake KO, Line PD, Grzyb K, Aamodt G, Aabakken L, Roset A, Hvinden AB, Bakka A, Eide J, Bjorneklett A, Vatn MH. Assessment of mucosal inflammation and blood flow in response to four weeks' intervention with probiotics in patients operated with a J-configurated ileal-pouch-anal-anastomosis (IPAA). Scand J Gastroenterol. 2004 Dec;39(12):1228-35. doi: 10.1080/00365520410009320. PMID 15743000
- [Background] Sharman MJ, Volek JS. Weight loss leads to reductions in inflammatory biomarkers after a very-low-carbohydrate diet and a low-fat diet in overweight men. Clin Sci (Lond). 2004 Oct;107(4):365-9. doi: 10.1042/CS20040111. PMID 15265001
- [Background] Middleton E Jr. Effect of plant flavonoids on immune and inflammatory cell function. Adv Exp Med Biol. 1998;439:175-82. doi: 10.1007/978-1-4615-5335-9_13. PMID 9781303
- [Background] McCarty MF. Low-insulin-response diets may decrease plasma C-reactive protein by influencing adipocyte function. Med Hypotheses. 2005;64(2):385-7. doi: 10.1016/j.mehy.2004.03.039. PMID 15607574
- [Background] De Caterina R, Liao JK, Libby P. Fatty acid modulation of endothelial activation. Am J Clin Nutr. 2000 Jan;71(1 Suppl):213S-23S. doi: 10.1093/ajcn/71.1.213S. PMID 10617974
- [Background] Giugliano D, Ceriello A, Esposito K. The effects of diet on inflammation: emphasis on the metabolic syndrome. J Am Coll Cardiol. 2006 Aug 15;48(4):677-85. doi: 10.1016/j.jacc.2006.03.052. Epub 2006 Jul 24. PMID 16904534
- [Background] Salehi-Abargouei A, Saraf-Bank S, Bellissimo N, Azadbakht L. Effects of non-soy legume consumption on C-reactive protein: a systematic review and meta-analysis. Nutrition. 2015 May;31(5):631-9. doi: 10.1016/j.nut.2014.10.018. Epub 2014 Nov 7. PMID 25837205
- [Background] Steckhan N, Hohmann CD, Kessler C, Dobos G, Michalsen A, Cramer H. Effects of different dietary approaches on inflammatory markers in patients with metabolic syndrome: A systematic review and meta-analysis. Nutrition. 2016 Mar;32(3):338-48. doi: 10.1016/j.nut.2015.09.010. Epub 2015 Oct 28. PMID 26706026
- [Background] Ahluwalia N, Andreeva VA, Kesse-Guyot E, Hercberg S. Dietary patterns, inflammation and the metabolic syndrome. Diabetes Metab. 2013 Apr;39(2):99-110. doi: 10.1016/j.diabet.2012.08.007. Epub 2012 Oct 11. PMID 23062863
- [Background] Berrino F, Bellati C, Secreto G, Camerini E, Pala V, Panico S, Allegro G, Kaaks R. Reducing bioavailable sex hormones through a comprehensive change in diet: the diet and androgens (DIANA) randomized trial. Cancer Epidemiol Biomarkers Prev. 2001 Jan;10(1):25-33. PMID 11205485
- [Background] Kaaks R, Bellati C, Venturelli E, Rinaldi S, Secreto G, Biessy C, Pala V, Sieri S, Berrino F. Effects of dietary intervention on IGF-I and IGF-binding proteins, and related alterations in sex steroid metabolism: the Diet and Androgens (DIANA) Randomised Trial. Eur J Clin Nutr. 2003 Sep;57(9):1079-88. doi: 10.1038/sj.ejcn.1601647. PMID 12947426
- [Background] Marlow G, Ellett S, Ferguson IR, Zhu S, Karunasinghe N, Jesuthasan AC, Han DY, Fraser AG, Ferguson LR. Transcriptomics to study the effect of a Mediterranean-inspired diet on inflammation in Crohn's disease patients. Hum Genomics. 2013 Nov 27;7(1):24. doi: 10.1186/1479-7364-7-24. PMID 24283712
- [Background] Browne RH. On the use of a pilot sample for sample size determination. Stat Med. 1995 Sep 15;14(17):1933-40. doi: 10.1002/sim.4780141709. PMID 8532986
- [Background] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782
- [Background] Pizzamiglio S, Cossa G, Gatti L, Beretta GL, Corna E, Tinelli S, Verderio P, Perego P. Simultaneous confidence intervals to compare gene expression profiles using ABC transporter TaqMan microfluidic cards. Oncol Rep. 2010 Mar;23(3):853-60. PMID 20127029
- [Background] Reid JF, Sokolova V, Zoni E, Lampis A, Pizzamiglio S, Bertan C, Zanutto S, Perrone F, Camerini T, Gallino G, Verderio P, Leo E, Pilotti S, Gariboldi M, Pierotti MA. miRNA profiling in colorectal cancer highlights miR-1 involvement in MET-dependent proliferation. Mol Cancer Res. 2012 Apr;10(4):504-15. doi: 10.1158/1541-7786.MCR-11-0342. Epub 2012 Feb 16. PMID 22343615
- [Background] Livak KJ, Schmittgen TD. Analysis of relative gene expression data using real-time quantitative PCR and the 2(-Delta Delta C(T)) Method. Methods. 2001 Dec;25(4):402-8. doi: 10.1006/meth.2001.1262. PMID 11846609
- [Derived] Illescas O, Ferrero G, Belfiore A, Pardini B, Tarallo S, Ciniselli CM, Noci S, Daveri E, Signoroni S, Cattaneo L, Mancini A, Morelli D, Milione M, Cordero F, Rivoltini L, Verderio P, Pasanisi P, Vitellaro M, Naccarati A, Gariboldi M. Modulation of faecal miRNAs highlights the preventive effects of a Mediterranean low-inflammatory dietary intervention. Clin Nutr. 2024 Apr;43(4):951-959. doi: 10.1016/j.clnu.2024.02.023. Epub 2024 Feb 26. PMID 38422953
- [Derived] Belfiore A, Ciniselli CM, Signoroni S, Gariboldi M, Mancini A, Rivoltini L, Morelli D, Masci E, Bruno E, Macciotta A, Ricci MT, Daveri E, Cattaneo L, Gargano G, Apolone G, Milione M, Verderio P, Pasanisi P, Vitellaro M. Preventive Anti-inflammatory Diet to Reduce Gastrointestinal Inflammation in Familial Adenomatous Polyposis Patients: A Prospective Pilot Study. Cancer Prev Res (Phila). 2021 Oct;14(10):963-972. doi: 10.1158/1940-6207.CAPR-21-0076. Epub 2021 Jul 12. PMID 34253565